CLINICAL TRIAL: NCT05968222
Title: Whole Body Vibration Exercise Intervention for Glycemic Control in Type 2 Diabetes Patients
Brief Title: Whole Body Vibration and Diabetes Type 2
Acronym: WBV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Vicente Rodríguez Pérez, Ph.D., University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Universidad de Salamanca
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Whole Body Vibration
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will undergo a determination of glycosylated hemoglobin, blood pressure, lipid profile, weight and height, as well as functional tests such as TUG, 10MWT, 5STS. Subsequently, they will be encouraged to continue their normal life insisting on the importance of glycemic controls before and after their daily physical exercise. In addition to continuing with the dietary measures recommended by their specialist.
- Experimental group (Experimental): Participants in the intervention group will be subjected to the following tests:
  * At the beginning of the intervention, a determination of glycosylated hemoglobin, blood pressure, lipid profile, weight, height and TUG, 10MWT, 5STS, which will be repeated after 12 weeks of intervention.
  * Before each training session, participants will undergo a basal blood glucose and blood pressure measurement, which will be repeated after the end of the session.
  * Each training session on the vibrating platform is composed of 6 exercises with a duration of 60 seconds with 60-second pauses between exercises and a warm-up exercise.
  Interventions: Other: Vibration exercise

INTERVENTIONS:
Other: Vibration exercise — Each training session on the vibrating platform is composed of 6 exercises with a duration of 60 seconds with 60-second pauses between exercises and a warm-up exercise
  Arms: Experimental group

SUMMARY:
Diabetes generates a great impact on society, as well as a concern for health professionals due to its high and increasing prevalence; there are more and more studies that demonstrate the effectiveness of vibration platforms and their benefits at a physiological level. The objective is to analyze the decrease in glycosylated hemoglobin and glycemia levels after the use of whole body vibration platforms and the possible inclusion of this therapeutic option within the usual treatments.The sample will be composed of people diagnosed with Type 2 Diabetes Mellitus in the Plasencia area (Cáceres, Extremadura). Participants will be randomly assigned to the intervention or control group using a randomization list and will follow the inclusion criteria: healthy type 2 diabetics between 50 and 60 years of age and not taking diabetes medication. All participants will undergo a determination of glycosylated hemoglobin, blood pressure, lipid profile, weight and height, and different functional tests such as TUG, 10MMT, 5STS. The experimental group will perform a full body vibration intervention on an oscillating platform for 12 weeks with a weekly frequency of 3 non-consecutive days and a duration of 12 minutes. The exercises will consist of 60 seconds of work and 60 seconds with rest. The control group will carry out their normal life insisting on the importance of glycemic controls before and after their daily physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Not taking medication for diabetes.

Exclusion Criteria:

* Suffer a pathology (such as diabetic retinopathy, diabetic nephropathy), mobility disability and/or comorbidities incompatible with physical exercise and the use of vibration platforms, previous hip or knee surgeries, cognitive impairment and neurological pathology

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c. | baseline and 12 weeks post
  HbA1c is a blood test to determine the average level of glucose or sugar in the blood during the last two or three months
Timed Up and Go 3 meters (TUG 3 m) | baseline and 12 weeks post
  The subject, seated with his back resting on the back of the chair (without armrests and height 43 cm), at the acoustic command following a five-second countdown, stands up, walks the expected distance, turns around a cone, goes back, turns 360° and sits down again. The test time stops when the subject returns to the starting position and is completely immobile.
10 Meters Walking Test (10 m) | baseline and 12 weeks post
  On command the subject covers the distance walking as fast as possible, without running.
Five times Sit To Stand (5STS) | baseline and 12 weeks post
  The subject, seated with his back supported on the chair (without armrests and height 43 cm), on command stands up and sits down five consecutive times, as fast as possible and without using the push of the hands on the quadriceps.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Spain

REFERENCES:
- [Background] Cardinale M, Bosco C. The use of vibration as an exercise intervention. Exerc Sport Sci Rev. 2003 Jan;31(1):3-7. doi: 10.1097/00003677-200301000-00002. PMID 12562163
- [Background] Rodriguez-Reyes RR, Navarro-Zarza JE, Tello-Divicino TL, Parra-Rojas I, Zaragoza-Garcia O, Guzman-Guzman IP. [Detection of cardiovascular risk in healthcare workers on the basis of WHO/JNC 7/ATP III criteria]. Rev Med Inst Mex Seguro Soc. 2017 May-Jun;55(3):300-308. Spanish. PMID 28440983
- [Background] del Pozo-Cruz B, Alfonso-Rosa RM, del Pozo-Cruz J, Sanudo B, Rogers ME. Effects of a 12-wk whole-body vibration based intervention to improve type 2 diabetes. Maturitas. 2014 Jan;77(1):52-8. doi: 10.1016/j.maturitas.2013.09.005. Epub 2013 Sep 18. PMID 24094494
- [Background] Bonaiuti D, Shea B, Iovine R, Negrini S, Robinson V, Kemper HC, Wells G, Tugwell P, Cranney A. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2002;(3):CD000333. doi: 10.1002/14651858.CD000333. PMID 12137611
- [Background] Behboudi L, Azarbayjani MA, Aghaalinejad H, Salavati M. Effects of aerobic exercise and whole body vibration on glycaemia control in type 2 diabetic males. Asian J Sports Med. 2011 Jun;2(2):83-90. doi: 10.5812/asjsm.34789. PMID 22375223
- [Background] Gusi N, Parraca JA, Olivares PR, Leal A, Adsuar JC. Tilt vibratory exercise and the dynamic balance in fibromyalgia: A randomized controlled trial. Arthritis Care Res (Hoboken). 2010 Aug;62(8):1072-8. doi: 10.1002/acr.20180. PMID 20235191
- [Background] Sanudo B, de Hoyo M, Carrasco L, McVeigh JG, Corral J, Cabeza R, Rodriguez C, Oliva A. The effect of 6-week exercise programme and whole body vibration on strength and quality of life in women with fibromyalgia: a randomised study. Clin Exp Rheumatol. 2010 Nov-Dec;28(6 Suppl 63):S40-5. Epub 2010 Dec 22. PMID 21122265
- [Background] Marazzi S, Kiper P, Palmer K, Agostini M, Turolla A. Effects of vibratory stimulation on balance and gait in Parkinson's disease: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2021 Apr;57(2):254-264. doi: 10.23736/S1973-9087.20.06099-2. Epub 2020 Jan 14. PMID 31939269
- [Background] Kang H, Lu J, Xu G. The effects of whole body vibration on muscle strength and functional mobility in persons with multiple sclerosis: A systematic review and meta-analysis. Mult Scler Relat Disord. 2016 May;7:1-7. doi: 10.1016/j.msard.2016.02.008. Epub 2016 Feb 8. PMID 27237747
- [Background] Slatkovska L, Alibhai SM, Beyene J, Hu H, Demaras A, Cheung AM. Effect of 12 months of whole-body vibration therapy on bone density and structure in postmenopausal women: a randomized trial. Ann Intern Med. 2011 Nov 15;155(10):668-79, W205. doi: 10.7326/0003-4819-155-10-201111150-00005. PMID 22084333
- [Background] Tseng CL, Brimacombe M, Xie M, Rajan M, Wang H, Kolassa J, Crystal S, Chen TC, Pogach L, Safford M. Seasonal patterns in monthly hemoglobin A1c values. Am J Epidemiol. 2005 Mar 15;161(6):565-74. doi: 10.1093/aje/kwi071. PMID 15746473